CLINICAL TRIAL: NCT06472245
Title: A Randomised, Open-label, Phase 3 Trial Comparing the Efficacy and Safety of OSE2101 Versus Docetaxel in HLA-A2 Positive Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC) With Secondary Resistance to Immune Checkpoint Inhibitor
Brief Title: Trial of Therapeutic Cancer Vaccine OSE2101 in Patients With Non-Small Cell Lung Cancer and Secondary Resistance to Immune Checkpoint Inhibitor
Acronym: ARTEMIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: OSE Immunotherapeutics (Industry)
Collaborators: Exystat (Other); Genome Diagnostics (GenDx) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSE2101C302
Record Dates: First submitted 2024-06-07; First posted 2024-06-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Patients With Non-Small Cell Lung Cancer
Keywords: Immune Checkpoint Inhibitor; Cancer vaccine; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Arm A: OSE2101 (Experimental): Unit dose: 1 mL corresponding to a total of 5 mg of the combination of peptides Mode/Route: Subcutaneous injection Regimen: One injection every three weeks for six cycles, then every eight weeks for the remainder of year one and, finally every twelve weeks until the end of second year.
  Interventions: Drug: OSE2101; Device: NGS HLAA2 assay
- Arm B: Docetaxel (Active Comparator): Unit dose: 75 mg/m2 Mode/Route: Intravenous infusion over 1 hour Regimen: One infusion every three weeks.
  Interventions: Drug: Docetaxel; Device: NGS HLAA2 assay
- GenDx CDx Tedopi (Other): System of qualitative companion diagnostic devices, consisting of a polymerase chain reaction (PCR) assay Amp-HLA-A-CDx Tedopi, a DNA library preparation assay, LFK-CDx Tedopi and the software NGSengine-CDx Tedopi.
  Interventions: Device: NGS HLAA2 assay

INTERVENTIONS:
Drug: OSE2101 — OSE2101 is a peptidic cancer vaccine composed of nine epitopes restricted to HLA-A2 phenotype targeting the tumor associated antigens of P53, HER-2, CEA, MAGE-2 and MAGE-3, and one pan-HLA DR binding epitope (PADRE), all epitopes emulsified in Montanide ISA 51TM adjuvant.
  Arms: Arm A: OSE2101
Drug: Docetaxel — Docetaxel is an antineoplastic agent that acts by disrupting the microtubular network in cells that is essential for mitotic and interphase cellular functions.
  Arms: Arm B: Docetaxel
Device: NGS HLAA2 assay — Amp-HLA-A-CDx Tedopi for amplification of human genomic DNA (gDNA), LFK-CDx Tedopi kit (library full kit) for library preparation, NGSengine-CDx Tedopi software for analysis of NGS data files.

SUMMARY:
Multicenter, randomized (2:1), open-label phase 3 study in HLA-A2 positive patients with squamous and non-squamous metastatic NSCLC with ICI secondary resistance.

Patients will be randomized into 2 arms (randomization 2:1): experimental Arm A with OSE2101 monotherapy or control Arm B SoC with docetaxel monotherapy. Stratification factors will be histology (squamous versus non squamous) and ECOG Performance Status (0 versus 1).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years
2. Patients expressing HLA-A2 phenotype in blood by pre-screening central laboratory
3. Patients with histologically or cytologically squamous or non-squamous documented NSCLC, metastatic stage at study entry, not eligible for definite surgery or radiation, without EGFR, ALK and ROS1 gene alterations eligible for targeted therapy; for patients with squamous NSCLC, the molecular tests are not mandatory if age ≥ 50 years old and smoker ≥ 15 pack years; other sensitizing mutations known to be immunosensitive are eligible in case of lack of local access to targeted therapy (i.e.; KRAS G12C and BRAF mutations) after Sponsor' agreement.
4. Patients with secondary resistance to ICI;

Other inclusion and exclusion criteria will apply per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
OS defined as time from randomization to death | From randomization date through study completion, an average of 3 years
  OS defined as time from randomization to death of any cause, censored until the data analysis cut-off date

CONTACTS AND LOCATIONS:
Locations (205):
- United States (79):
  - Clinical Research Advisors, LLC, Beverly Hills, California
  - Clinical Research Advisors - Encino, Encino, California
  - Clinical Research Advisors - West Hollywood, Los Angeles, California
  - Clinical Research Advisors - Korea Town, Los Angeles, California
  - SCL Health - Saint Joseph Hospital Cancer Center, Littleton, Colorado
  - Lutheran Medical Center - Cancer Centers of Colorado, Wheat Ridge, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Comprehensive Hematology Oncology - Bradenton Clinic, Bradenton, Florida
  - Comprehensive Hematology Oncology - Brandon Clinic, Brandon, Florida
  - Cancer Specialists of North Florida - Fleming Island, Fleming Island, Florida
  - Cancer Specialists of North Florida - Riverside, Jacksonville, Florida
  - Cancer Specialists of North Florida Southside, Jacksonville, Florida
  - Cancer Specialists of North Florida - Northside, Jacksonville, Florida
  - Cancer Specialists of North Florida - Southpoint, Jacksonville, Florida
  - Cancer Specialists of North Florida - Baptist South, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville Beach, Florida
  - Comprehensive Hematology Oncology - Largo Clinic, Largo, Florida
  - Cancer Specialists of North Florida - Beaches, Neptune Beach, Florida
  - Comprehensive Hematology Oncology - Palm Harbor Clinic, Palm Harbor, Florida
  - Cancer Specialists Of North Florida - St. Augustine, Saint Augustine, Florida
  - Comprehensive Hematology Oncology - Bayfront Clinic, St. Petersburg, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - Comprehensive Hematology Oncology - Trinity Clinic, Trinity, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Alliance for Multispecialty Research (AMR) - Kansas City Oncology, Merriam, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Pontchartrain Cancer Center - Covington Office, Covington, Louisiana
  - Pontchartrain Cancer Center - Hammond Office, Hammond, Louisiana
  - Ascension Saint Agnes Hospital, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Nebraska Hematology-Oncology - Revive Research Institute LLC, Lincoln, Nebraska
  - New York Cancer & Blood Specialists - Babylon Medical Oncology, Babylon, New York
  - Optum Medical Care - Carmel/Brewster Campus, Brewster, New York
  - Brooklyn Radiation Oncology, Brooklyn, New York
  - Optum Medical Care - Fishkill Westage Campus, Fishkill, New York
  - Clinical Research Alliance, Lake Success, New York
  - Optum Medical Care - Mount Kisco Campus 90, Mount Kisco, New York
  - New York Cancer & Blood Specialists - New Hyde Park, New Hyde Park, New York
  - Optum Hematology Oncology - Lake Success, New Hyde Park, New York
  - New York Cancer & Blood Specialists - Cancer Center - Research Headquarters, New York, New York
  - New York Cancer & Blood Specialists - Central Park Medical Oncology, New York, New York
  - New York Cancer & Blood Specialists - Patchogue Medical Oncology, Patchogue, New York
  - New York Cancer & Blood Specialists - Port Jefferson Medical Oncology, Port Jefferson Station, New York
  - New York Cancer & Blood Specialists - Port Jefferson Station Medical Oncology, Port Jefferson Station, New York
  - Optum Medical Care - Poughkeepsie, Poughkeepsie, New York
  - New York Cancer & Blood Specialists - Eastchester Cancer Care Center, The Bronx, New York
  - New York Cancer & Blood Specialists - Riverhead Medical Oncology, The Bronx, New York
  - Mercy Health - Perrysburg Cancer Center, Perrysburg, Ohio
  - Mercy Health - St. Anne Cancer Center, Toledo, Ohio
  - Bon Secours Hematology and Oncology, Greenville, South Carolina
  - Tennessee Oncology - Chattanooga - Medical Park II, Chattanooga, Tennessee
  - Tennessee Oncology - Chattanooga - Downtown, Chattanooga, Tennessee
  - Tennessee Oncology - Chattanooga - GHCR Site I, Chattanooga, Tennessee
  - Tennessee Oncology - Chattanooga - Memorial Plaza, Chattanooga, Tennessee
  - Tennessee Oncology - Cleveland Clinic, Cleveland, Tennessee
  - Tennessee Oncology - Cookeville Clinic, Cookeville, Tennessee
  - Tennessee Oncology - Dickson Clinic, Dickson, Tennessee
  - Tennessee Oncology - Franklin Clinic, Franklin, Tennessee
  - Tennessee Oncology - Gallatin Clinic, Gallatin, Tennessee
  - Tennessee Oncology - Hendersonville Clinic, Hendersonville, Tennessee
  - Tennessee Oncology - Hermitage - Summit Clinic, Hermitage, Tennessee
  - Tennessee Oncology - Lebanon Clinic, Lebanon, Tennessee
  - Tennessee Oncology - Murfreesboro Clinic, Murfreesboro, Tennessee
  - Tennessee Oncology - Nashville - Centennial Center for Blood Cancers Clinic, Nashville, Tennessee
  - Tennessee Oncology - Nashville - Centennial Clinic - Medical Oncology, Nashville, Tennessee
  - Tennessee Oncology - Nashville - Midtown Center for Blood Cancers, Nashville, Tennessee
  - Tennessee Oncology - Nashville - St. Thomas Midtown Clinic, Nashville, Tennessee
  - Tennessee Oncology - Nashville - St. Thomas West Clinic, Nashville, Tennessee
  - Tennessee Oncology - Nashville - Skyline Clinic, Nashville, Tennessee
  - Tennessee Oncology - Nashville - Southern Hills Clinic, Nashville, Tennessee
  - Greco-Hainsworth Tennessee Oncology Centers for Research (GHCR) - Corporate, Nashville, Tennessee
  - Tennessee Oncology - Shelbyville Clinic, Shelbyville, Tennessee
  - Tennessee Oncology - Smyrna Clinic, Smyrna, Tennessee
  - Northwest Medical Specialties - Bonney Lake, Bonney Lake, Washington
  - Northwest Medical Specialties - Federal Way, Federal Way, Washington
  - Northwest Medical Specialties - Gig Harbor, Gig Harbor, Washington
  - Northwest Medical Specialties - Puyallup Medical Oncology, Puyallup, Washington
  - Northwest Medical Specialties - Tacoma, Tacoma, Washington
- Belgium (9):
  - Algemeen Ziekenhuis Klina, Brasschaat, Antwerpen
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt, Limburg
  - Algemeen Ziekenhuis Maria Middelares, Ghent, Oost-Vlaaderen
  - Centre Hospitalier Universitaire Université Catholique de Louvain Namur - Site Sainte-Elisabeth, Namur, Wallonia
  - Algemeen Ziekenhuis Groeninge - Campus Kennedylaan, Kortrijk, West-Vlaanderen
  - Algemeen Ziekenhuis Delta - Campus Rembert Torhout, Roeselare, West-Vlaanderen
  - Algemeen Ziekenhuis Delta - Campus Rumbeke, Roeselare, West-Vlaanderen
  - Algemeen Ziekenhuis Delta - Campus Menen, Roeselare, West-Vlaanderen
- Canada (3):
  - Centre Intégré Universitaire de Santé et de Services Sociaux du Saguenay - Lac-Saint-Jean, Chicoutimi, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Intégré de Santé et de Services Sociaux du Bas-Saint-Laurent, Rimouski, Quebec
- France (29):
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon, Alpes-de-Haute-Provence
  - Nouvel Hôpital Civil, Strasbourg, Alsace
  - Hôpital Louis Pradel, Bron, Auvergne-Rhône-Alpes
  - Centre Hospitalier Lyon-Sud, Lyon, Auvergne-Rhône-Alpes
  - Hôpital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes
  - Institut Paoli-Calmettes, Marseille, Bouches-du-Rhône
  - Centre Hospitalier Régional et Universitaire de Besançon - Hôpital Jean-Minjoz, Besançon, Doubs
  - Centre Hospitalier Regional Universitaire Brest - Hopital de la Cavale Blanche, Brest, Finistère
  - Hôpital Emile Muller, Mulhouse, Grand Est
  - Centre Hospitalier Universitaire Dupuytren 1, Limoges, Haute-Vienne
  - Hôpital Arnaud de Villeneuve, Montpellier, Hérault
  - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Institut de Cancérologie de l'Ouest - Saint-Herblain - Site René Gauducheau, Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier (Ch) De Cholet, Cholet, Maine-et-Loire
  - Hôpital Larrey, Toulouse, Midi-pyrenees
  - Hôpital Nord de Marseille, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Côte Basque, Bayonne, Pyrénées-Atlantiques
  - Hôpital Michallon, La Tronche, Rhône
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Institut Sainte Catherine, Avignon, Vaucluse
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Universitaire De Nantes - Hôpital Nord Laennec, Nantes
  - Hôpital Avicenne, Bobigny, Île-de-France Region
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Île-de-France Region
  - Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region
  - Hôpital Cochin, Paris, Île-de-France Region
  - Hôpital Tenon, Paris, Île-de-France Region
- Germany (12):
  - Thoraxklinik-Heidelberg, Heidelberg, Baden-Wurttemberg
  - Robert-Bosch-Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Asklepios Fachkliniken München-Gauting, Gauting, Bavaria
  - München Klinik Bogenhausen, München, Bavaria
  - Klinikum Kassel, Kassel, Hesse
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Gießen und Marburg - Gießen, Homburg, Saarland
  - Krankenhaus Martha-Maria Halle-Dölau, Halle, Saxony-Anhalt
  - LungenClinic Grosshansdorf, Großhansdorf, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin, Berlin
- Greece (11):
  - Metropolitan Hospital, Piraeus, Athens
  - Saint Savvas Anticancer - Oncological Hospital of Athens, Athens, Attica
  - Henry Dunant Hospital Center, Athens, Attica
  - General Hospital for Thoracic Diseases Sotiria, Athens, Attica
  - Agii Anargiri Cancer Hospital, Nea Kifissia, Attica
  - Clinic Agios Loukas, Thessaloniki, Central Macedonia
  - University General Hospital of Heraklion (PAGNI), Heraklion, Crete
  - General Hospital of Thessaloniki Papageorgiou, Thessaloniki, Macedoni
  - University General Hospital of Patras, Patra, Peloponnese
  - Theagenio Anti-Cancer Hospital of Thessaloniki, Thessaloniki, Thessaloniki
  - University General Hospital of Larissa, Larissa, Thessaly
- Hungary (3):
  - Mátrai Gyógyintézet, Gyöngyös, Heves County
  - Országos Korányi Pulmonológiai Intézet, Budapest
  - Clinexpert Kft. telephelye, Bugát Pál Kórház - Phase I. Clinical Trial Site, Gyöngyös
- Italy (17):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola, Forlì-Cesena
  - Presidio Ospedaliero di Lucca, San Filippo, Lucca
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Istituto Clinico Humanitas, Rozzano, Milan
  - Azienda Ospedaliera Universitaria - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Naples
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Ospedale P. Pederzoli - Casa di Cura Privata S.p.A., Legnago, Verona
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale Policlinico San Martino, Genova
  - Ospedale Vito Fazzi Lecce, Lecce
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Ospedale Busonera - Istituto Oncologico Veneto (IOV) - Padua, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda Unità Sanitaria Locale della Romagna - Ospedale Infermi di Rimini, Rimini
  - IRCCS Istituto Nazionale Tumori Regina Elena, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - Azienda Ospedaliera Universitaria Senese - L'ospedale Santa Maria alle Scotte, Siena
- Netherlands (3):
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen, Groningen
- Poland (6):
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin, Greater Poland Voivodeship
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeylandów, Poznan, Greater Poland Voivodeship
  - Centrum Onkologii Im. Prof. F. Łukaszczyka w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Lódzkie
  - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk, Pomeranian Voivodeship
- Portugal (5):
  - Unidade Local de Saúde de Coimbra, Coimbra
  - Hospital CUF Descobertas, Lisbon
  - Unidade Local de Saúde de Santa Maria, E. P. E. - Hospital Pulido Valente, Lisbon
  - Hospital CUF Porto, Porto
  - Unidade Local de Saúde de Gaia/Espinho, E. P. E, Vila Nova de Gaia
- Romania (3):
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca, Cluj
  - Centrul de Oncologie Sf Nectarie, Craiova, Dolj
  - SC OncoMed SRL, Timișoara, Timiș County
- Spain (20):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), L'Hospitalet de Llobregat, Barcelona
  - Biocruces Bizkaia Instituto de Investigación Sanitaria, Barakaldo, Biscay
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - HC Marbella, Marbella, Malaga
  - Clínica Mi Tres Torres, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (5):
  - University Hospitals of Leicester NHS Trust, Leicester, England
  - The Christie NHS Foundation Trust, Manchester, England
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral, England
  - The Royal Marsden NHS Foundation Trust, Sutton, England
  - NHS Grampian, Aberdeen, Scotland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Besse B, Felip E, Garcia Campelo R, Cobo M, Mascaux C, Madroszyk A, Cappuzzo F, Hilgers W, Romano G, Denis F, Viteri S, Debieuvre D, Galetta D, Baldini E, Razaq M, Robinet G, Maio M, Delmonte A, Roch B, Masson P, Schuette W, Zer A, Remon J, Costantini D, Vasseur B, Dziadziuszko R, Giaccone G; ATALANTE-1 study group. Randomized open-label controlled study of cancer vaccine OSE2101 versus chemotherapy in HLA-A2-positive patients with advanced non-small-cell lung cancer with resistance to immunotherapy: ATALANTE-1. Ann Oncol. 2023 Oct;34(10):920-933. doi: 10.1016/j.annonc.2023.07.006. Epub 2023 Sep 11. PMID 37704166